CLINICAL TRIAL: NCT03457298
Title: Lateral Ridge Augmentation Using a Volume Maintaining Collagen Scaffold (Ossix Volumax) Versus Freeze-dried Bone Allograft (FDBA) With Collagen Membrane
Brief Title: Lateral Ridge Augmentation Using a Volume Maintaining Collagen Scaffold Versus Allograft With Collagen Membrane.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0014-18-RMB CTIL
Record Dates: First submitted 2018-02-26; First posted 2018-03-07 (Actual); Last update posted 2019-05-20 (Actual); Status verified 2019-05

CONDITIONS: Alveolar Ridge Augmentation, Dental Implants

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ossix Volumax (Experimental): lateral bone augmentation using volume maintaining collagen scaffold (Ossix Volumax)
  Interventions: Device: Ossix Volumax
- FDBA with collagen membrane (Active Comparator): lateral bone augmentation using the current gold standard FDBA plus resorbable collagen membrane
  Interventions: Device: FDBA with collagen membrane

INTERVENTIONS:
Device: Ossix Volumax — Ossix Volumax is intended to be used for Lateral ridge augmentation
  Arms: Ossix Volumax
Device: FDBA with collagen membrane — freeze-dried bone allograft (FDBA) with collagen membrane
  Arms: FDBA with collagen membrane

SUMMARY:
The aim of the current study is to compare lateral bone augmentation using the current gold standard (FDBA plus resorbable collagen membrane) versus Ossix Volumax as a stand-alone material.

DETAILED DESCRIPTION:
One of the major problems in implant therapy is the need to regenerate bone after its resorption because of periodontal disease, traumatic extraction or surgical removal associated with treatment of invasive lesions.

Ossix Volumax is a novel volume maintaining collagen scaffold designed for bone augmentation in the atrophic ridge. It is 1-2 mm in thickness and undergoes mineralization progressing into ossification.

Thirty subjects requiring lateral bone augmentation of the maxilla or the mandible will be recruited study: Of these, twenty will be recruited and treated at the School of Dental Medicine, Harvard University, Boston, USA and ten (10) at the School of Graduate Dentistry, Rambam health care campus, Haifa, Israel.

Hypothesis:

The use of Ossix Volumax as a stand-alone augmentation material will results similar increase in the ridge width and volume compared to FDBA and barrier membrane when coupled together.

ELIGIBILITY:
Inclusion Criteria:

1. Patients age 18 to 85 years of age.
2. Alveolar ridge atrophy (<5 mm) in the horizontal dimension requiring bone augmentation.
3. Implant therapy is scheduled for this site.
4. Willing to participate in the study and follow all the post-op visits.

Exclusion Criteria:

1. Systemic condition requiring prophylactic antibiotics.
2. The Introduction( I.V.) use of medication related osteonecrosis of the jaw ( MRONJ) or the use of such medication Per Os (P.O.) for five or more years, patients with at least three month drug holiday with a C-terminal cross-linking telopeptide (CTX) > 150 pg/ml are eligible.
3. The use of medication known to impair healing (clinician desecration).
4. Unable to place implant for whatever reason.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-11-07 (Actual); Primary Completion 2020-04 (Estimated); Study Completion 2020-07 (Estimated)

PRIMARY OUTCOMES:
Changes in socket width mm | baseline( prior to augmentation) and 9 months (implant placement)
  Clinical measurement of the ridge width as -2, -5 & -8 mm from crest at the Region of interest (ROI) using a caliper

SECONDARY OUTCOMES:
Changes in Ridge height mm | baseline( prior to augmentation) and 9 months (implant placement)
  Ridge height from a pre-determined landmark using a 15mm Dental probe

CONTACTS AND LOCATIONS:
Overall Officials: Eli Machtei, DMD, Principal Investigator — Rambam Health Care Campus
Locations (1):
- Rambam Health Care Campus, Dept. of Periodontology, Haifa, Israel